CLINICAL TRIAL: NCT06489639
Title: School-based Treatment of Social Anxiety: A Randomized and Controlled Study Using Developmentally Oriented Cognitive Therapy for Social Anxiety Disorder
Brief Title: School-based Treatment of Social Anxiety With Developmentally Oriented Cognitive Therapy for Social Anxiety Disorder
Acronym: SBT-DOCT-SAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Klaus Ranta (Other)
Collaborators: University of Helsinki (Other); Finnish Institute for Health and Welfare (Other Government); University of Eastern Finland (Other)
Responsible Party: Sponsor-Investigator, Klaus Ranta, Associate Professor, Tampere University
Organization: Tampere University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R22123
Record Dates: First submitted 2024-06-28; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Social Anxiety Disorder; Social Anxiety; Adolescent - Emotional Problem
Keywords: social anxiety, adolescents, cognitive behavioural therapy
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Developmentally Oriented Cognitive Therapy for Social Anxiety Disorder (DOCT-SAD) (Experimental): Developmentally Oriented Cognitive Therapy for Social Anxiety Disorder (DOCT-SAD) is a ten-session, combined group/individual intervention program for treating social anxiety and social anxiety disorder in adolescents. It consists of four individual and six group sessions delivered during a ten-week period. The number of adolescents in each DOCT-SAD group varies between four and six. One or both parents attend two of the individual DOCT-SAD sessions.
  Interventions: Behavioral: DOCT-SAD
- Standard Counseling (SC) (Active Comparator): Standard Counseling (SC) is an intervention consisting of counseling sessions delivered by a school health and welfare (SHWS) professional (i.e., school nurse, school social worker, or school psychologist) to support a student with social anxiety. The defined length of intervention is ten weeks. In SC, routine professional working methods and procedures available to the SHWS professional delivering the intervention are used.
  Interventions: Behavioral: SC

INTERVENTIONS:
Behavioral: DOCT-SAD — Developmentally Oriented Cognitive Therapy for Social Anxiety Disorder is a 10-session, combined individual/group clinical intervention for treating social anxiety in adolescents. It consists of four individual and six group sessions during ten weeks. DOCT-SAD groups are formed for 4-6 adolescnts. One parent or both parents attend two of the individual sessions.
  Other Names: Developmentally Oriented Cognitive Therapy for Social Anxiety Disorder
  Arms: Developmentally Oriented Cognitive Therapy for Social Anxiety Disorder (DOCT-SAD)
Behavioral: SC — Standard Counseling (SC) is a intervention consisting of counseling sessions delivered by a school health and welfare (SHWS) professional (i.e., school nurse, school social worker, or school psychologist) to support a student with social anxiety. The defined length of intervention is ten weeks, and number of sessions will be according to what is routinely agreed between the professional and the adolescent. In SC, routine professional working methods and procedures available to the SHWS professional delivering the intervention are used.
  Other Names: Standard Counseling
  Arms: Standard Counseling (SC)

SUMMARY:
The goal of this randomized controlled trial is to find out whether the brief, 10-session Developmentally Oriented Cognitive Therapy for Social Anxiety Disorder (DOCT-SAD) is more effective than standard counseling (SC) to treat Social Anxiety Disorder (SAD) among 12 to 17-year-old adolescents with SAD.

Potential participants for the study are identified from school health and well-being services (SHWS). The DOCT-SAD is delivered by method-trained school psychologists working in the SHWS. SC will be provided by non-method-trained SHWS professionals (i.e. school nurses, social workers or school psychologists) according to their routine counselling practice.

The main research questions of the study are:

1. Is DOCT-SAD more effective than SC for alleviating symptoms of social anxiety?
2. Is DOCT-SAD more effective than SC to produce diagnostic remission from primary SAD and alleviating symptom severity associated with SAD?
3. Is DOCT-SAD more effective than SC for alleviating co-occurring depressive symptoms, interference in daily functioning due to worry or fears, and for increasing general well-being, positive mental health, and for improving the quality of life among adolescents with SAD?

Researchers will compare DOCT-SAD with SC to see if DOCT-SAD is effective in the treatment of SAD in adolescents.

Participants will:

* be treated either with DOCT-SAD or SC for 10 weeks.
* be followed up and assessed clinically at six-month and twelve-month follow-up points.

DETAILED DESCRIPTION:
Aim:

The aim of this randomized controlled trial is to investigate whether a brief, 10-session intervention, the Developmentally Oriented Cognitive Therapy for Social Anxiety Disorder (DOCT-SAD; in Finnish Tosi minä -treeni) is more effective than standard counseling (SC) for alleviating symptoms of social anxiety and to treat Social Anxiety Disorder (SAD) among adolescents identified from School Health and Well-being Services (SHWS) of mandatory public schools.

Participants:

Participants comprise of students in the grades 7-9 of the public secondary schools, and students in the 1st or 2nd year-course of public high schools and vocational schools in the Tampere area of Finland. They are aged from 12 to 17 years. All participants will present with primary SAD according to DSM-5 criteria. In total, 156 students will be recruited.

Procedure:

Participants are identified by professionals working in the School Health and Welfare Services (SHWS). Recruitment is enhanced by sending information on social anxiety, SAD and the research project to all SHWS professionals of the participating schools using e-mails, online meetings, and pre-recorded online presentations. In addition, families of students in the participating schools are approached with brief informative leaflets about social anxiety and the study via e-mail. Potential participants for the trial will be identified in the schools using a two-stage screening and detection procedure in the SHWS and a SAD detection toolkit.

In the first stage, adolescents with suspected social anxiety are evaluated by SHWS professionals (i.e., school nurses, school social workers and school psychologists) from their current student clients or from their new encounters with students using the SAD detection toolkit. The detection toolkit consists of: 1. symptom measure of social anxiety (SPIN) with instructions on scoring and the clinical cutoff; 2. treatment suitability evaluation checklist consisting of inclusion/exclusion criteria for the study in an abbreviated form, and 3. pictorially enhanced one-page psychoeducation leaflet designed to help in the differentiation between core symptoms of anxiety and depression, and differentiating between different types of anxiety.

In the second stage, the DOCT-SAD-trained school psychologists, who also have been trained in diagnostic evaluation of SAD, act as consultants for other SHWS professionals. Once contacted by non-trained SHWS professional they discuss with them and review all information gathered. The either confrirm or reject a likely diagnosis of primary SAD. These DOCT-trained school psychologists refer the eligble students to the clinical research interview.

The clinical intake interview:

The clinicical research team evaluates the referred adolescents and assigns clinical diagnoses according DSM-5. The ADIS-5 interview schedule is used for diagnostic assessment of anxiety disorders, and the associated CSR scale for is used to assess the severity of SAD and other anxiety disorders. The K-SADS-PL interview schedule usis used for the diagnostic assessment of other DSM-5 disorders. Subjects who present with primary SAD are asked to participate, and adolescents and their parents who give their written content are taken in to the study.

Randomization:

After intake to the study subjects will be randomized to intervention group (i.e., to receive DOCT-SAD delivered by the school psychologists) or to comparison group (i.e., to receive SC provided by a SHWS professional according to her/his routine professional practice). For DOCT -SAD between 4 and 6 adolescents are recruited to each group randomization is performed during the school term when enough referrals.

Delivery of interventions:

The DOCT-SAD will be delivered by method-trained and weekly supervised school psychologists working in the SHWSs. SC will be provided by non-trained SHWS professionals (i.e. either school nurses, social workers or psychologists) according their routine counselling practice. The school psychologists delivering the DOCT-SAD receive weekly, group-based method supervision.

DOCT-SAD:

The DOCT-SAD is a combined individual/group, ten-session intervention for social anxiety treatment largely based largely on the cognitive therapy program CT-SAD, developed in the University of Oxford, UK. It has been modified and theoretically expanded to address the features and challenges unique to the developmental phase of adolescence. DOCT-SAD consists of four indidual and six group sessions. Parents attend two of the sessions. DOCT-SAD uses the main treatment components from the DOCT-SAD program, derived from the cognitive model of SAD by David M. Clark and Adrian Wells in 1995. These componenets include psychoeducation of SAD, individual/historical symptom formulation according to cognitive model, experiential exercise on the consequences of engaging in safety behaviours, attention training, repeated behavioural experiments, dropping of safety behaviours, imagery rescripting on traumatic memories, and cognitive work on beliefs.

Added theoretical sources of DOCT-SAD include use of the theoretical model of core fears of social anxiety disorder being related to experienced flaws/deficiencies in the self as presented by David Moscovitch in 2009. The development of a acceptable, positive self-identity is seen essential for adolescents, and DOCT-SAD program makes use of original materials instuting therapist and adolescents to work on restructuring dysfunctional thoughts and emotions related to social anxiety in the context of experienced self-image/self-concept. Another theoretical influence is drawn from the reseach on psychotherapeutic use of of self-compassion as an antidote to self-cricism, as developed by Paul Gilbert in 2009, and applied to treatment of social anxiety by Lynne Henderson and colleagues in 2014.

In DOCT-SAD programme emphasis on developmental factors is reflected in the combined individual / group format of the treatment. Positive peer modeling and peer support are encouraged in the group. DOCT-SAD materials are developmentally informed, with much emphasis given to normalization of anxiety, normative fears of being deviant in the eyes of peers, need for being accepted and the normative high priority given to peer opinion. Group and pair exercices and out-of-office behavioural experiments are planned to encourage adolescents to practice abandoning their safety behaviors based on what they believe other people consider acceptable. Brief modules to develop self-compassion are included. As process, adolescents work in DOCT-SAD to progress from negative self-experience, self-criticism and self-concealment to being all the more their authentic self, and lastly to being their authentic self and simultaneously being self-supportive in anxiety inducing social situations. An empahsis is given to finding associations between adolescents' SAD symptoms and their self-experience and perceived flaws and deficiencies in their their self-experience. Repeated pair, group and field practice of dropping of self-concealment as a safety behaviour is performed using behavioral experiments and self-exposuresand home work assignments.

SC:

Standard Counseling (SC) is an intervention consisting of counseling sessions delivered by a school health and welfare (SHWS) professional (i.e., school nurse, school social worker, or school psychologist) to support a student with social anxiety. The defined length of intervention is ten weeks. In SC, routine professional working methods and procedures available to the SHWS professional delivering the intervention are used in the counseling.

In addition to methods, number of sessions, treatment goals, and possible involvement of parents are agreed between the counselor, adolescent and parent in the same way as they are routinely agreed by the SHWS professional in her/his work with the students.

Thus, SC represents an intervention that is routinely delivered by a SHWS professional with a student with social anxiety.

Evaluation of outcomes:

The design of this trial is randomized, controlled trial. Participants in both intervention arms are evaluated prior to treatment, at post-treatment (2,5 months), and at 6-month and 12-month follow-up points aftter the intervention with the same methods and measures.

Clinical change:

Both self-report instuments (SPIN, SAFE, PHQ-9, CALIS-C, CALIS-P, YP-CORE, SWEMWBS, WHOQOL-BREF) and clinical interviews (ADIS-5, with associated CSR scale, K-SADS-PL) are used for assessing clinical change.

Feasibility of DOCT-SAD and SC:

Feasibility of both DOCT-SAD and SC as interventions for the participants, for their parents, and for the professionals delivering the interventions is evaluated after both interventions using a structured interview schedule.

Economic evaluation and additional service use:

An economic evaluation of DOCT-SAD and SC includes an assessment of professionals' time resource allocated for the intervention during the ten weeks, and an evaluation of additional service use of the particpiants in both intervention groups. The professionals delivering DOCT-SAD and SC are interviewed on the total time they have allocated to the intervention using a structured questonnaire. Participants' use of additional (i.e., other than DOCT-SAD or SC) healthcare and counseling services during past six months are evaluated twice: first at the intake interview for the study and for the second time at 12-month follow-up point. A structured survey form is used to collect the service use data.

ELIGIBILITY:
Inclusion criteria:

* age 13-17 years
* diagnosis of DSM-5 SAD (Social Anxiety Disorder)
* SAD is the primary mental health disorder
* motivation of the adolescent and parent to attend DOCT-SAD / SC as described in the study protocol
* good command of the Finnish language.

Exclusion criteria:

* intellectual deficit
* presence of primary autism spectrum disorder
* marked psychotic symptoms or psyhotic disorder
* severe eating disorder, depression or primary other anxiety disorder requiring acute treatment which need to be prioritized above treatment of social anxiety
* acute suicidality or suicide risk
* substance use or substance use disorder requiring child protection measures
* presence of contextual/environmental risk factors in the participants surroundings which require child protection measures

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 156 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-reported social anxiety symptoms | From treatment startpoint to treatment endpoint (2,5 months), to 6-month follow-up point, and to 12-month follow-up point
  Change in self-reported social anxiety symptoms assessed with the Social Phobia Inventory (SPIN)
Diagnostic status of SAD | From treatment startpoint to treatment endpoint (2,5 months), to 6-month follow-up point, and to 12-month follow-up point
  Change in the diagnostic status of SAD according DSM-5 criteria, assessed with ADIS-5 interview schedule
Clinical severity of SAD symptoms | From treatment startpoint to treatment endpoint (2,5 months), to 6-month follow-up, and to 12-month follow-up
  Change in the clinical severity of SAD symptoms assessed with the CSR scale of the ADIS-5 interview schedule

SECONDARY OUTCOMES:
Self-reported safety behaviours associated with SAD | From treatment startpoint to treatment endpoint (2,5 months), to 6-month follow-up, and to 12-month follow-up
  Change in self-reported safety behaviours associated with SAD assessed with the Subtle Avoidance Frequency Examination (SAFE)
Self-reported depressive symptoms | From treatment startpoint to treatment endpoint (2,5 months), to 6-month follow-up, and to 12-month follow-up
  Change in self-reported depressive symptoms assessed with the Patient Health Questionnaire-9 (PHQ-9)
Self-reported life interference due to fears and worries | From treatment startpoint to treatment endpoint (2,5 months), to 6-month follow-up, and to 12-month follow-up
  Change in self-reported life inteference due to fears and worries assessed with the Child Anxiety Life Interference Scale (CALIS-C)
Parent-reported life interference due to adolescent's fears and worries | From treatment startpoint to treatment endpoint (2,5 months), to 6-month follow-up, and to 12-month follow-up
  Change in parent-reported life inteference due to adolescent's fears and worries assessed with the Child Anxiety Life Interference Scale for Parents (CALIS-P)
Self-reported general well-being | From treatment startpoint to treatment endpoint (2,5 months), to 6-month follow-up, and to 12-month follow-up
  Change in self-reported general well-being assessed with the Young Person's Clinical Outcomes in Routine Evaluation (YP-CORE)
Self-reported positive mental health | From treatment startpoint to the end of the follow-up period (12 months)
  Change in self-reported positive mental health assessed with the Short version of the Warwick-Edinburgh Mental Well-being Scale (SWEMWBS)
Self-reported quality of life | From treatment startpoint to the end of the follow-up period (12 months)
  Change in self-reported quality of life assessed with the World Health Organization Quality of Life -BREF (WHOQOL-BREF)

OTHER OUTCOMES:
Use of healthcare and consulting services during prior six months | From treatment startpoint to the end of the follow-up period (12 months)
  Change in adolescent's use of healthcare and consulting services during prior six months reported by the adolescent and parents, assessed with a structured survey form

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Ranta, MD, PhD, Study Director — Tampere University
Locations (1):
- Tampere University, Tampere, Pirkanmaa, Finland